CLINICAL TRIAL: NCT05511194
Title: Safety and Efficacy of Enhanced Recovery After Surgery Therapeutic Protocol for Complicated Appendicitis in Children
Brief Title: Safety and Efficacy of ERAS Therapeutic Protocol for Complicated Appendicitis in Children
Acronym: ERAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, CLOTILDE FUENTES OROZCO, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F-2022-1302-028
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Enhanced Recovery After Surgery; Appendicitis; Children, Only
Keywords: Enhanced Recovery After Surgery; Appendicitis complicated; Appendectomy; Children; Perioperative period
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial, single blind.
Who Masked: Participant
Masking Description: The patient will be assigned to a control group or an experimental group based on simple random probabilistic sampling, using software (OxMaR: Oxford Minimization and Randomization, 2019) for minimization and randomization of clinical studies, single blind. A different postoperative treatment scheme will be applied for each of the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group: scheduled nausea and vomiting prophylaxis the first postoperative 24 hours, start liquid diet 8 hours postoperative, if tolerated, advance to a soft diet in the next shift, double IV antibiotic scheme (ceftriaxone, metronidazole) for at least 3 days and change to oral route upon discharge to complete 10 days of antibiotics, discharge upon accomplish discharge criteria (at least 3 days with IV antibiotic scheme, tolerance to feeding, tolerance to postoperative pain and 24 hours without the presence of fever).
  Interventions: Other: Enhanced Recovery After Surgery therapeutic protocol
- Control Group (Other): Control Group: use of antiemetic only in case of nausea or vomiting, start of liquid diet when presenting intestinal transit data (channeling of gases or presence of evacuation), if they tolerate advancing to a soft diet in the next shift, triple IV antibiotic regimen (ampicillin, amikacin, metronidazole) for at least 5 days and change to oral route upon discharge to complete 10 days of antibiotics, discharge upon accomplish discharge criteria (at least 5 days with IV antibiotic regimen, tolerance to feeding, tolerance to postoperative pain and 24 hours without the presence of fever).
  Interventions: Other: Conventional management

INTERVENTIONS:
Other: Enhanced Recovery After Surgery therapeutic protocol — Feeding and early ambulation, double short IV antibiotic regimen.
  Arms: Experimental Group
Other: Conventional management — Delayed feeding and ambulation, triple short IV antibiotic regimen.
  Arms: Control Group

SUMMARY:
Complicated appendicitis in pediatrics is frequent, potentially serious and complex to manage. The implementation of a ERAS model would allow optimizing perioperative care, offering a shorter hospital stay, reducing complications associated with medical care and costs, although adequate multidisciplinary management is necessary. The objective of the study is to evaluate the safety and efficacy of the application of a ERAS therapeutic protocol and compare them with the safety and efficacy of conventional management in children with complicated appendicitis.

DETAILED DESCRIPTION:
1. All patients who meet the indicated criteria will be included, including signing an informed consent in the immediate postoperative period, and will be assigned to a control group or an experimental group based on simple random probabilistic sampling, using software (OxMaR: Oxford Minimization and Randomization, 2019) for minimization and randomization of clinical studies, single blind. A different postoperative treatment scheme will be applied for each of the groups.
2. Post-surgical indications for each group:

   For both groups: assisted ambulation when recovering from the anesthetic effect, surgical wound care (daily bathing and cleaning the wound with soap and water, dressing change every 24 hours or as needed), preferably non-opioid analgesics.

   Experimental Group: scheduled nausea and vomiting prophylaxis the first postoperative 24 hours, start liquid diet 8 hours postoperative, if tolerated, advance to a soft diet in the next shift, double IV antibiotic scheme (ceftriaxone, metronidazole) for at least 3 days and change to oral route upon discharge to complete 10 days of antibiotics, discharge upon accomplish discharge criteria (at least 3 days with IV antibiotic scheme, tolerance to feeding, tolerance to postoperative pain and 24 hours without the presence of fever).

   Control Group: use of antiemetic only in case of nausea or vomiting, start of liquid diet when presenting intestinal transit data (channeling of gases or presence of evacuation), if they tolerate advancing to a soft diet in the next shift, triple IV antibiotic regimen (ampicillin, amikacin, metronidazole) for at least 5 days and change to oral route upon discharge to complete 10 days of antibiotics, discharge upon accomplish discharge criteria (at least 5 days with IV antibiotic regimen, tolerance to feeding, tolerance to postoperative pain and 24 hours without the presence of fever).
3. The information on each case will be recorded on a data collection sheet, that will include an identification sheet (number of patient, telephone number, age and sex), date of admission, conditions at the time of admission, weight and height to calculate nutritional status, time of evolution in hours of the clinical picture until admission to the operating room, if he received antibiotic treatment prior to admission, post-surgical diagnosis (appendicitis phase), anesthetic method used, type of analgesic used, antibiotic scheme used, date of discharge and complications at discharge.
4. Outpatient follow-up will be carried out with control at 7, 15 and 30 postoperative days, in person to identify the presence of complications through questioning and physical examination, as well as histopathological diagnosis review. These data will also be recorded on the collection sheet.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 1 and 17, who underwent surgery at the UMAE Hospital de Pediatría CMNO and who at the time of surgery are determined to be in a gangrenous or perforated phase.

Exclusion Criteria:

* Patients who, prior to surgery, present symptoms of intestinal obstruction, abdominal sepsis, or suffer from any underlying disease.
* Patients who require placement of a nasogastric tube or abdominal drainage during the intervention.
* Patients who were operated in another unit and enter the service for follow-up.
* Patients whose legal guardians do not agree to sign consent to participate in the protocol.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Hospitalary stay | 120 days
  Days elapsed between the admission of the patient for in-hospital management and his discharge by medical decision. Care effectiveness indicator.
Complications | 120 days
  Adverse events presented as a consequence of the evolution of a disease or a medical intervention. Indicator of safety of the intervention carried out.

SECONDARY OUTCOMES:
Hospital costs | 120 days
  Costs based on unit costs by level of medical care (Official Gazette of the Federation).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Ambriz, MD, Study Director — UMAE Pediatric Hospital CMNO IMSS

IPD SHARING:
Plan to Share IPD: No
Not required

REFERENCES:
- [Result] Omling E, Salo M, Saluja S, Bergbrant S, Olsson L, Persson A, Bjork J, Hagander L. Nationwide study of appendicitis in children. Br J Surg. 2019 Nov;106(12):1623-1631. doi: 10.1002/bjs.11298. Epub 2019 Aug 6. PMID 31386195
- [Result] Addiss DG, Shaffer N, Fowler BS, Tauxe RV. The epidemiology of appendicitis and appendectomy in the United States. Am J Epidemiol. 1990 Nov;132(5):910-25. doi: 10.1093/oxfordjournals.aje.a115734. PMID 2239906
- [Result] Garst GC, Moore EE, Banerjee MN, Leopold DK, Burlew CC, Bensard DD, Biffl WL, Barnett CC, Johnson JL, Sauaia A. Acute appendicitis: a disease severity score for the acute care surgeon. J Trauma Acute Care Surg. 2013 Jan;74(1):32-6. doi: 10.1097/TA.0b013e318278934a. PMID 23271074
- [Result] Bhangu A, Soreide K, Di Saverio S, Assarsson JH, Drake FT. Acute appendicitis: modern understanding of pathogenesis, diagnosis, and management. Lancet. 2015 Sep 26;386(10000):1278-1287. doi: 10.1016/S0140-6736(15)00275-5. PMID 26460662
- [Result] Bonadio W, Rebillot K, Ukwuoma O, Saracino C, Iskhakov A. Management of Pediatric Perforated Appendicitis: Comparing Outcomes Using Early Appendectomy Versus Solely Medical Management. Pediatr Infect Dis J. 2017 Oct;36(10):937-941. doi: 10.1097/INF.0000000000001025. PMID 26669739
- [Result] Bolmers MD, van Rossem CC, Gorter RR, Bemelman WA, van Geloven AAW, Heij HA; Snapshot Appendicitis Collaborative Study group. Imaging in pediatric appendicitis is key to a low normal appendix percentage: a national audit on the outcome of appendectomy for appendicitis in children. Pediatr Surg Int. 2018 May;34(5):543-551. doi: 10.1007/s00383-018-4244-2. Epub 2018 Mar 9. PMID 29523946
- [Result] Fujishiro J, Watanabe E, Hirahara N, Terui K, Tomita H, Ishimaru T, Miyata H. Laparoscopic Versus Open Appendectomy for Acute Appendicitis in Children: a Nationwide Retrospective Study on Postoperative Outcomes. J Gastrointest Surg. 2021 Apr;25(4):1036-1044. doi: 10.1007/s11605-020-04544-3. Epub 2020 Mar 3. PMID 32128682
- [Result] Knaapen M, van Amstel P, van Amstel T, The SML, Bakx R, van Heurn ELWE, Gorter RR. Outcomes after appendectomy in children with acute appendicitis treated at a tertiary paediatric centre: results from a retrospective cohort study. Langenbecks Arch Surg. 2021 Feb;406(1):163-169. doi: 10.1007/s00423-020-01976-y. Epub 2020 Aug 28. PMID 32860108
- [Result] Martinez-Perez A, Paya-Llorente C, Santarrufina-Martinez S, Sebastian-Tomas JC, Martinez-Lopez E, de'Angelis N. Predictors for prolonged length of stay after laparoscopic appendectomy for complicated acute appendicitis in adults. Surg Endosc. 2021 Jul;35(7):3628-3635. doi: 10.1007/s00464-020-07841-9. Epub 2020 Aug 7. PMID 32767147
- [Result] Howell EC, Dubina ED, Lee SL. Perforation risk in pediatric appendicitis: assessment and management. Pediatric Health Med Ther. 2018 Oct 26;9:135-145. doi: 10.2147/PHMT.S155302. eCollection 2018. PMID 30464677
- [Result] Zavras N, Vaos G. Management of complicated acute appendicitis in children: Still an existing controversy. World J Gastrointest Surg. 2020 Apr 27;12(4):129-137. doi: 10.4240/wjgs.v12.i4.129. PMID 32426092
- [Result] Zani A, Hall NJ, Rahman A, Morini F, Pini Prato A, Friedmacher F, Koivusalo A, van Heurn E, Pierro A. European Paediatric Surgeons' Association Survey on the Management of Pediatric Appendicitis. Eur J Pediatr Surg. 2019 Feb;29(1):53-61. doi: 10.1055/s-0038-1668139. Epub 2018 Aug 15. PMID 30112745
- [Result] Yousef Y, Youssef F, Homsy M, Dinh T, Pandya K, Stagg H, Baird R, Laberge JM, Poenaru D, Puligandla P, Shaw K, Emil S. Standardization of care for pediatric perforated appendicitis improves outcomes. J Pediatr Surg. 2017 Dec;52(12):1916-1920. doi: 10.1016/j.jpedsurg.2017.08.054. Epub 2017 Sep 5. PMID 28935397
- [Result] Lam JY, Beaudry P, Simms BA, Brindle ME. Impact of implementing a fast-track protocol and standardized guideline for the management of pediatric appendicitis. Can J Surg. 2021 Jul 5;64(4):E364-E370. doi: 10.1503/cjs.005420. PMID 34223740
- [Result] Do-Wyeld M, Cundy TP, Court-Kowalski S, Dandie L, Cooper C, Burgoyne L, Cooksey R, Khurana S. Improving quality and efficiency of care for advanced appendicitis in children. ANZ J Surg. 2021 Jul;91(7-8):1497-1503. doi: 10.1111/ans.16929. Epub 2021 May 20. PMID 34013543
- [Result] Wilmore DW, Kehlet H. Management of patients in fast track surgery. BMJ. 2001 Feb 24;322(7284):473-6. doi: 10.1136/bmj.322.7284.473. No abstract available. PMID 11222424
- [Result] Taurchini M, Del Naja C, Tancredi A. Enhanced Recovery After Surgery: a patient centered process. J Vis Surg. 2018 Feb 27;4:40. doi: 10.21037/jovs.2018.01.20. eCollection 2018. PMID 29552522
- [Result] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Result] Kehlet H. [Fast-track surgery: the facts and the challenges]. Cir Esp. 2006 Oct;80(4):187-8. doi: 10.1016/s0009-739x(06)70955-1. No abstract available. Spanish. PMID 17040666
- [Result] Kehlet H. Fast-track surgery-an update on physiological care principles to enhance recovery. Langenbecks Arch Surg. 2011 Jun;396(5):585-90. doi: 10.1007/s00423-011-0790-y. Epub 2011 Apr 6. PMID 21468643
- [Result] Brindle ME, Heiss K, Scott MJ, Herndon CA, Ljungqvist O, Koyle MA; on behalf Pediatric ERAS (Enhanced Recovery After Surgery) Society. Embracing change: the era for pediatric ERAS is here. Pediatr Surg Int. 2019 Jun;35(6):631-634. doi: 10.1007/s00383-019-04476-3. Epub 2019 Apr 25. PMID 31025092
- [Result] Kehlet H, Wilmore DW. Fast-track surgery. Br J Surg. 2005 Jan;92(1):3-4. doi: 10.1002/bjs.4841. No abstract available. PMID 15635603
- [Result] Roberts K, Brindle M, McLuckie D. Enhanced recovery after surgery in paediatrics: a review of the literature. BJA Educ. 2020 Jul;20(7):235-241. doi: 10.1016/j.bjae.2020.03.004. Epub 2020 May 6. No abstract available. PMID 33456956
- [Result] Bailey K, Choynowski M, Kabir SMU, Lawler J, Badrin A, Sugrue M. Meta-analysis of unplanned readmission to hospital post-appendectomy: an opportunity for a new benchmark. ANZ J Surg. 2019 Nov;89(11):1386-1391. doi: 10.1111/ans.15362. Epub 2019 Jul 30. PMID 31364257
- [Result] Hajibandeh S, Hajibandeh S, Bill V, Satyadas T. Meta-analysis of Enhanced Recovery After Surgery (ERAS) Protocols in Emergency Abdominal Surgery. World J Surg. 2020 May;44(5):1336-1348. doi: 10.1007/s00268-019-05357-5. PMID 31897698
- [Result] Sazhin AV, Nechay TV, Titkova SM, Tyagunov AE, Anurov MV, Melnikov-Makarchuk KY, Tyagunov AA, Ermakov IV, Glagolev NS, Kurashinova LS, Ivanova EA, Nechay VS, Karpov AV, Mirzoyan AT, Ivakhov GB, Balakirev YS. [Comparison of standard and fast track rehabilitation in patients with acute appendicitis. Intermediate results of multicenter prospective randomized trial]. Khirurgiia (Mosk). 2018;(9):15-23. doi: 10.17116/hirurgia2018090115. Russian. PMID 30307416
- [Result] Trejo-Avila ME, Romero-Loera S, Cardenas-Lailson E, Blas-Franco M, Delano-Alonso R, Valenzuela-Salazar C, Moreno-Portillo M. Enhanced recovery after surgery protocol allows ambulatory laparoscopic appendectomy in uncomplicated acute appendicitis: a prospective, randomized trial. Surg Endosc. 2019 Feb;33(2):429-436. doi: 10.1007/s00464-018-6315-9. Epub 2018 Jul 9. PMID 29987566
- [Result] Trejo-Avila M, Cardenas-Lailson E, Valenzuela-Salazar C, Herrera-Esquivel J, Moreno-Portillo M. Ambulatory versus conventional laparoscopic appendectomy: a systematic review and meta-analysis. Int J Colorectal Dis. 2019 Aug;34(8):1359-1368. doi: 10.1007/s00384-019-03341-y. Epub 2019 Jul 5. PMID 31273450
- [Result] Tlacuilo-Parra A, Lopez-Valenzuela SP, Ambriz-Gonzalez G, Guevara-Gutierrez E. [Seguridad y eficacia del modelo de atencion fast-track vs. atencion convencional en apendicitis no complicada del paciente pediatrico]. Cir Cir. 2018;86(5):412-416. doi: 10.24875/CIRU.18000189. Spanish. PMID 30226494
- [Result] Yu YR, Smith CM, Ceyanes KK, Naik-Mathuria BJ, Shah SR, Vogel AM, Carberry KE, Nuchtern JG, Lopez ME. A prospective same day discharge protocol for pediatric appendicitis: Adding value to a common surgical condition. J Pediatr Surg. 2017 Oct 9:S0022-3468(17)30633-4. doi: 10.1016/j.jpedsurg.2017.10.011. Online ahead of print. PMID 29103787
- [Result] Frazee R, Abernathy S, Davis M, Isbell T, Regner J, Smith R. Fast track pathway for perforated appendicitis. Am J Surg. 2017 Apr;213(4):739-741. doi: 10.1016/j.amjsurg.2016.08.006. Epub 2016 Oct 20. PMID 27816201
- [Result] Shbat L, Emil S, Elkady S, Baird R, Laberge JM, Puligandla P, Shaw K. Benefits of an abridged antibiotic protocol for treatment of gangrenous appendicitis. J Pediatr Surg. 2014 Dec;49(12):1723-5. doi: 10.1016/j.jpedsurg.2014.09.039. Epub 2014 Oct 11. PMID 25487469
- [Result] Lasso Betancor CE, Ruiz Hierro C, Vargas Cruz V, Orti Rodriguez RJ, Vazquez Rueda F, Paredes Esteban RM. [Implementation of "fast-track" treatment in paediatric complicated appendicitis]. Cir Pediatr. 2013 Apr;26(2):63-8. Spanish. PMID 24228355
- See also: 17. Malaekah H, Makhdoom F, Almedbal H and Aggarwal R. Acute Appendicitis Pathways: A Systemic Review. Surgical Science, 2021; 12: 143-159. — https://www.scirp.org/journal/paperinformation.aspx?paperid=109433